CLINICAL TRIAL: NCT03978039
Title: The "BCB-sarcomes" Database: the Database of the French Sarcoma Group Dedicated to the Collection of Clinical and Biological Data for All Sarcomas
Brief Title: National Clinical and Biological Sarcoma Database : An Initiative of the French Sarcoma Group
Acronym: BCB-Sarcomes
Status: Recruiting | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: French Sarcoma Group (Other)
Responsible Party: Sponsor
Other Study IDs: IB2012-BCB-SARCOMES
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Sarcoma
Keywords: patterns of care; access to care; survival; experts' network
MeSH Terms: conditions — Sarcoma | interventions — Drug Therapy; Adjuvants, Immunologic; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with sarcoma: Patients with a sarcoma diagnosed in a French Comprehensive cancer Center
  Interventions: Drug: Chemotherapy; Drug: Immunotherapeutic Agent; Drug: target treatment; Procedure: Surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Chemotherapy — treatment as per standard of care
Drug: Immunotherapeutic Agent — treatment as per standard of care
Drug: target treatment — treatment as per standard of care
Procedure: Surgery — treatment as per standard of care
Radiation: Radiotherapy — treatment as per standard of care

SUMMARY:
The BCB SARCOMES database is a clinical and biological national database dedicated to sarcoma that contains 3 main databases with specific aims: the first is the pathology database (French expert network dedicated to the management of bone sarcomas [RESOS] / French expert network dedicated to the pathology of sarcomas [RREPS]), dedicated to systematic review of mesenchymal tumor diagnostics nationwide; the second is clinical (RESOS / French expert clinical network for sarcomas [NETSARC]), collecting multidisciplinary tumor boards (MDTB) data of patients nationwide, and the third (CONTICABASE / BONE / GIST) is dedicated to collecting patients longitudinal/follow up data, with a focus on treatments of every events, and a catalogue of associated samples.

Primary objectives of BCB-SARCOMES are the following: description of the patterns of care and treatment outcomes, assessment of the prognostic factors of patients' outcomes.

With the financial support of the French National Cancer Institute [Institut National du cancer [INCa]).

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of sarcoma
* Diagnosis in a French Comprehensive Cancer Center
* Any age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to next treatment (TNT) | 2 years
  Time from the systemic treatment onset to the next treatment or death due to any cause, whichever comes first. When neither death nor new systemic therapy is observed, TNT is censored at the date of last patient contact.
Time to next treatment (TNT) | 5 years
  Time from the systemic treatment onset to the next treatment or death due to any cause, whichever comes first. When neither death nor new systemic therapy is observed, TNT is censored at the date of last patient contact.
Overall survival (OS) | 2 years
  Interval between diagnosis and the time of death. When death is not observed, OS is censored at the date of last patient contact.
Overall survival (OS) | 5 years
  Interval between diagnosis and the time of death. When death is not observed, OS is censored at the date of last patient contact.

CONTACTS AND LOCATIONS:
Overall Officials: Maud Toulmonde, MD, Study Chair — Institut Bergonié, Bordeaux, France; Axel Le Cesne, MD/PhD, Study Chair — Institut Gustave Roussy, Villejuif, France; Jean-Yves Blay, MD/PhD, Study Chair — Centre Léon Bérard, Lyon, France
Locations (3):
- France (3):
  - Institut Bergonié, Comprehensive Cancer Center, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Comprehensive Cancer Center, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Savina M, Le Cesne A, Blay JY, Ray-Coquard I, Mir O, Toulmonde M, Cousin S, Terrier P, Ranchere-Vince D, Meeus P, Stoeckle E, Honore C, Sargos P, Sunyach MP, Le Pechoux C, Giraud A, Bellera C, Le Loarer F, Italiano A. Patterns of care and outcomes of patients with METAstatic soft tissue SARComa in a real-life setting: the METASARC observational study. BMC Med. 2017 Apr 10;15(1):78. doi: 10.1186/s12916-017-0831-7. PMID 28391775
- [Background] Toulmonde M, Bonvalot S, Meeus P, Stoeckle E, Riou O, Isambert N, Bompas E, Jafari M, Delcambre-Lair C, Saada E, Le Cesne A, Le Pechoux C, Blay JY, Piperno-Neumann S, Chevreau C, Bay JO, Brouste V, Terrier P, Ranchere-Vince D, Neuville A, Italiano A; French Sarcoma Group. Retroperitoneal sarcomas: patterns of care at diagnosis, prognostic factors and focus on main histological subtypes: a multicenter analysis of the French Sarcoma Group. Ann Oncol. 2014 Mar;25(3):735-742. doi: 10.1093/annonc/mdt577. PMID 24567518
- [Background] Blay JY, Soibinet P, Penel N, Bompas E, Duffaud F, Stoeckle E, Mir O, Adam J, Chevreau C, Bonvalot S, Rios M, Kerbrat P, Cupissol D, Anract P, Gouin F, Kurtz JE, Lebbe C, Isambert N, Bertucci F, Toumonde M, Thyss A, Piperno-Neumann S, Dubray-Longeras P, Meeus P, Ducimetiere F, Giraud A, Coindre JM, Ray-Coquard I, Italiano A, Le Cesne A. Improved survival using specialized multidisciplinary board in sarcoma patients. Ann Oncol. 2017 Nov 1;28(11):2852-2859. doi: 10.1093/annonc/mdx484. PMID 29117335
- See also: Related Info — https://conticabase.sarcomabcb.org/